CLINICAL TRIAL: NCT01878370
Title: Optimizing Audit and Feedback for Primary Care - Testing Scalable Approaches to Providing Feedback Reports, a Cluster-randomized Trial
Brief Title: Audit and Feedback for Primary Care: a Cluster-randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Institute for Clinical Evaluative Sciences (Other); Canadian Institutes of Health Research (CIHR) (Other Government); Heart and Stroke Foundation of Canada (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 075-2013
Record Dates: First submitted 2013-06-12; First posted 2013-06-14 (Estimated); Last update posted 2014-11-24 (Estimated); Status verified 2014-11

CONDITIONS: Diabetes; Hypertension; Ischemic Heart Disease
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Myocardial Ischemia | interventions — Practice Guidelines as Topic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High risk (Experimental): Feedback reports focusing on the identification and management of patients who appear to have poorly managed diseases and who may require recall into clinic.
  Interventions: Other: High risk
- Best Practice (Experimental): Feedback reports focusing on the achievement of optimal care targets for patients with chronic disease.
  Interventions: Other: Best Practice

INTERVENTIONS:
Other: High risk — Aggregate-level feedback reports focusing on the proportion of patients with hypertension and/or diabetes and/or ischemic heart disease meeting criteria for high-risk sent via courier every six months and available on a password protected website. Family physicians in this arm will also have access through this website to a list of chart numbers identifying those patients at highest risk.
  Family physicians in Arm 2 are asked to complete a worksheet that also includes goal setting and action planning, but focuses on reducing the number of patients with high-risk criteria and offers some suggested practice-based approaches.
  Arms: High risk
Other: Best Practice — Standard, aggregate-level feedback reports focusing on the proportion of patients with hypertension and/or diabetes and/or ischemic heart disease meeting targets sent via courier every six months and available on a password protected website. Family physicians in this arm will also have access through this website to patient-level data to identify patients not achieving optimal quality of care targets.
  Family physicians in Arm 1 are asked to complete a worksheet that follows continuous quality improvement principles, including setting an aim statement, engagement with team members in the clinic, testing change concepts at first on a small scale, and then scaling up in a effort to spread best practices.
  Arms: Best Practice

SUMMARY:
In a previous study, the investigators delivered graphs to family physicians that outlined the proportion of patients with a history of diabetes or heart disease achieving evidence-based quality targets derived from guideline recommendations. A qualitative evaluation found that participating family physicians did not act upon the feedback for two main reasons. First, they felt that targets recommended in guidelines often did not apply for particular patients. Second, they complained that had difficulty using the feedback reports that only provided aggregate level data for clinical action. In this cluster-randomized trial, the investigators test two approaches to conducting audit and feedback that aims to address these issues. The investigators hypothesize that feedback identifying a small number of patients at high-risk for cardiovascular events requiring action will more effectively lead to changes in clinical behavior than feedback identifying all patients not reaching optimal care targets.

DETAILED DESCRIPTION:
For the last two years, all physicians contributing data to the Electronic Medical Record Administrative data Linked Database (EMRALD) have received two feedback reports. The first focused on diabetes and the second on patients with heart disease. The reports provide aggregate information regarding the proportion of the family physician's patients meeting quality targets, but no patient-specific information. Currently the feedback is sent to physicians by courier from the EMRALD team every six months.

The intervention arms in this trial are as follows:

* Arm 1 - Standard, aggregate-level feedback reports focusing on the proportion of patients with hypertension and/or diabetes and/or ischemic heart disease meeting targets sent via courier every six months and available on a password protected website. Family physicians in this arm will also have access through this website to patient-level data to identify patients not achieving optimal quality of care targets.
* Arm 2 - Aggregate-level feedback reports focusing on the proportion of patients with hypertension and/or diabetes and/or ischemic heart disease meeting criteria for high-risk sent via courier every six months and available on a password protected website. Family physicians in this arm will also have access through this website to a list of chart numbers identifying those patients at highest risk.

Both arms will have the opportunity to receive continuing medical education credits by completing worksheets that prompt them to reflect upon the data. Family physicians in Arm 1 are asked to complete a worksheet that follows continuous quality improvement principles, including setting an aim statement, engagement with team members in the clinic, testing change concepts at first on a small scale, and then scaling up in a effort to spread best practices. Family physicians in Arm 2 are asked to complete a worksheet that also includes goal setting and action planning, but focuses on reducing the number of patients with high-risk criteria and offers some suggested practice-based approaches.

ELIGIBILITY:
Inclusion Criteria:

* Family physicians belonging to and sharing data with the Electronic Medical Record Administrative Linked Database in Ontario
* Patients rostered to these family physicians with diabetes or hypertension or ischemic heart disease

Exclusion Criteria:

* Family physicians without at least two years of Electronic Medical Record data in EMRALD
* Family physicians without at least 100 rostered, active patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 177 (Actual)
Dates: Start 2013-06; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
composite quality score | 12 months
  The number of best-practice quality indicators that a patient is achieving divided by the number for which they are eligible.
composite high risk score | 12 months
  The number of high risk indicators a patient meets divided by the number for which they are eligible.
Proportion of patients with perfect composite quality score | 12 months
  perfect composite quality score is equal to one hundred percent
Proportion of patients with perfect composite high risk score | 12 months
  perfect composite high risk score is zero

SECONDARY OUTCOMES:
Blood pressure | 12 months
cholesterol (LDL) | 12 months

OTHER OUTCOMES:
Each metric within the composite scores | 12 months
  For Hypertension (HTN):
  Blood Pressure (BP) tested in 15 months (M) BP meeting target BP test in 4 M if >target Weight (WT) measured in 15 M Lipids measures in 15 M
  For Diabetes:
  HbA1c tested in 6 M HbA1c < 7 BP <130/80 Angiotensin agent (ACE/ARB) if also HTN WT measured within 15 M Lipids in 15 M LDL <2 Statin if >50yrs Albumin-creatinine ratio in 15 M
  For Heart disease:
  BP in 15 M BP meeting target Anti-platelet (or Anti-coagulant) WT within 15 M Lipids measured within 15 M LDL <2 Statin
  For Diabetes High Risk:
  no HbA1c 15 M HbA1c >9 no BP in 15 M BP >160/100 no ACE/ARB if also HTN no WT within 24 M no lipids measured within 36 M LDL >4
  For Heart disease high risk:
  no BP in 24 M BP >160/100 no anti-platelet (anti-coagulant) no WT within 24 M no lipids measured within 36 M LDL >4
  For Hypertension high risk:
  no BP in 24 M BP >160/100 no WT within 24 M no lipids in 36 M

CONTACTS AND LOCATIONS:
Overall Officials: Karen Tu, MD MSc, Principal Investigator — Institute for Clinical Evaluative Sciences
Locations (1):
- Institute for Clinical Evaluative Sciences, Toronto, Ontario, Canada